CLINICAL TRIAL: NCT07167732
Title: Dragonfly Study: An International, Prospective, Longitudinal, Observational Natural History Study of Children and Adults Living With CTNNB1 Neurodevelopmental Syndrome
Brief Title: CTNNB1 Neurodevelopmental Syndrome - Natural History Study
Acronym: Dragonfly
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: The University of New South Wales (Other); University of Ljubljana School of Medicine, Slovenia (Other); CTNNB1 Foundation (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Assoc. Prof. Damjan Osredkar, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-174/2024-2711-8; J7-4537 (Other Grant/Funding Number: Slovenian Research And Innovation Agency)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: CTNNB1 Neurodevelopmental Syndrome
Keywords: CTNNB1 neurodevelopmental syndrome; Natural History Study; CTNNB1 gene mutation; Autism Spectrum Disorder; Beta-catenin; Developmental Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities | interventions — Neurologic Examination; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Venepuncture will be performed by a qualified member of the research team on all participants at each visit and 2x 5ml of blood will be collected (< 0.8 ml/kg) for analysis of DNA methylation and RNA expression, and analysis of serum for neurofilaments, b-catenin, and zinc. All blood samples will be labelled with the study ID and visit number and processed at the laboratory of the UMCL following the protocol "CTNNB1".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and Adults with CTNNB1 Neurodevelopmental Syndrome
  Interventions: Diagnostic Test: A General Medical and Neurological Assessment; Diagnostic Test: World Health Organisation (WHO) Motor Milestones; Diagnostic Test: Burke-Fahn-Marsden Dystonia Rating Scale; Diagnostic Test: Spastic Paraplegia Rating Scale; Diagnostic Test: 5. CTNNB1-Related Neurodevelopmental Disorder (NEDSDV) Cardiac Health Questionnaire; Diagnostic Test: 10m Walk-Run Test; Diagnostic Test: The Nine Hole Peg Test; Diagnostic Test: The Gross Motor Function Classification System; Diagnostic Test: Bayley Scales of Infant and Toddler Development-4: Fine Motor, Gross Motor, Language, and Cognitive Scales; Diagnostic Test: Wechsler Non-Verbal Scale of Ability; Diagnostic Test: The Vineland Adaptive Behaviour Scales - 3; Diagnostic Test: Aberrant Behaviour Checklist -Community; Diagnostic Test: The Modified Checklist for Autism in Toddlers; Diagnostic Test: The Autism Spectrum Quotient Questionnaire -Children's Version; Diagnostic Test: The Autism-Spectrum Quotient (AQ)-Adolescent Version; Diagnostic Test: Continuous Movement Monitoring (Actimyo/Syde); Diagnostic Test: Sleep Disturbance Scale for Children; Diagnostic Test: Seizure Diary; Diagnostic Test: 30min EEG Recording; Diagnostic Test: PedsQL Family Impact Module; Diagnostic Test: PedsQL Core Module; Diagnostic Test: Blood Sample Collection; Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: A General Medical and Neurological Assessment — Clinical assessments will consist of gathering demographic data, detailed relevant medical history, and parents' perspectives on treatment priorities, clinical trial interest, and acceptability of risk in future clinical trials. A general medical and neurological examination will be performed by a trained and skilled physician with a valid Good Clinical Practice Certification.
Diagnostic Test: World Health Organisation (WHO) Motor Milestones — Ages of six WHO Motor milestones achievements - sitting without support, hands and knees crawling, standing with support, walking with support, standing independently, and walking independently - will be assessed. The age of milestone achievement will be compared to normative variations in age as recommended by the WHO (WHO, 2006).
Diagnostic Test: Burke-Fahn-Marsden Dystonia Rating Scale — The Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS; Burke, Fahn, Marsden et. al, 1985) is a universally applied biomarker for the severity of dystonia in children and adults. The scale consists of a movement and disability subscale (Burke-Fahn-Marsden Movement Scale [BFMMS] and Burke-Fahn-Marsden Disability Scale [BFMDS], respectively. Only the BFMMS will be assessed. The BFMMS measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs) with scores ranging from 0 (minimum) to 120 (maximum).
Diagnostic Test: Spastic Paraplegia Rating Scale — The Spastic Paraplegia Rating Scale (SPRS; Schüle et al., 2006) is a 13-item scale used to measure disease severity in spastic paraplegia. The items include walking distance without pause, gait quality, maximum gait speed, climbing stars, arising from chair, spasticity of hip adductor and knee flexion muscles, weakness of hip abduction and foot dorsiflexion, contracture of lower limbs, pain related to spasticity, and bladder and bowel function. Each item has a score ranging from 0 to 4, where 0 represents no dysfunction and 4 represents most severe dysfunction. The score result is calculated by adding single scores of each of the 13 items. The total score varies between 0 (no dysfunction) and 52 (most severe dysfunction).
Diagnostic Test: 5. CTNNB1-Related Neurodevelopmental Disorder (NEDSDV) Cardiac Health Questionnaire — In a recent study (Sinibaldi et al., 2023), several patients with NEDSDV showed heart abnormalities. To expand on that, investigators developed a parent report questionnaire on the presence of potential heart defects.
Diagnostic Test: 10m Walk-Run Test — The 10m Walk-Run Test is is a performance measure used to assess walking or gait speed in meters per second over a short distance. It involves measuring the time it takes for a person to walk the distance, with results reported in meters/second (m/s). The patient's ability to walk at both comfortable and fast speeds can be measured, and assistive devices can be used. The test will be performed in ambulant children by an experienced physiotherapist.
Diagnostic Test: The Nine Hole Peg Test — The Nine-Hole Peg Test (9-HPT; Kellor et al., 1971) is a standardized, quantitative assessment used to measure finger dexterity. It is administered by asking the client to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. The 9-HPT has been validated for children above the age of 4 years (Poole et al., 2006). The test will be performed in children over 4 years old by a trained investigator.
Diagnostic Test: The Gross Motor Function Classification System — The Gross Motor Function Classification System (GMFCS; Palisano, Rosenbaum, Bartlett, Livingston, 2007) is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy on the basis of their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility. Distinctions between levels are based on functional abilities, the need for assistive technology, including hand-held mobility devices (walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement. The questionnaire is available for four age groups of children and youth: 2 to < 4 years, 4 to < 6 years, 6 to < 12 years, and 12 to 18 years.
Diagnostic Test: Bayley Scales of Infant and Toddler Development-4: Fine Motor, Gross Motor, Language, and Cognitive Scales — Bayley Scales of Infant and Toddler Development-4 (BSID-4; Bayley et al., 2019) is an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood. It consists of 419 items across 5 scales, each of which can be administered separately - Cognitive Scale (81 items), Language Scale (79 items), Motor Scale (104 items), Social-Emotional Scale (35 items), and Adaptive Behavior Scale (120 items). In our study, Motor, Language and Cognitive scales will be performed by a trained psychologist - if possible, at the patient's home country and in their native language.
Diagnostic Test: Wechsler Non-Verbal Scale of Ability — Wechsler Nonverbal Scale of Ability (WNV, Wechsler et al., 2006) is a standardized, individually administered test designed to assess general cognitive ability in individuals aged 4 to 21 years, particularly those who may have language, cultural, or communication challenges that make traditional verbal IQ tests less appropriate. It consists of six different subtests that are utilized based on the participant's age. In our study, the test will be performed in children above the age of 4 years by a trained psychologist - if possible, at the patient's home country and in their native language.
Diagnostic Test: The Vineland Adaptive Behaviour Scales - 3 — The Vineland Adaptive Behaviour Scales (VABS-3; Sparrow et al., 2018) is a standardized assessment tool that utilizes semi-structured interview to measure adaptive behaviour and support the diagnosis of intellectual and developmental disabilities, autism, and developmental delays. It is validated for children of all ages and consists of five primary domains (Communication, Daily Living Skills, Socialization, Motor Skills, and Adaptive Behavior Composit).
Diagnostic Test: Aberrant Behaviour Checklist -Community — The Aberrant Behaviour Checklist-Community (ABC-C) is a parent report behavioural rating scale designed to assess problem behaviours in individuals with developmental disabilities. It consists of 58 likert-type items across five domains (Irritability, Social Withdrawal, Stereotypic Behaviour, Hyperactivity, and Inappropriate Speech) with responses ranging from "not at all a problem" to "the problem is severe in degree".
Diagnostic Test: The Modified Checklist for Autism in Toddlers — The Modified Checklist for Autism in Toddlers (M-CHAT; Robins, Fein, & Barton, 2009) is a 2-stage parent report screening tool to assess risk for autism spectrum disorder (ASD). It is validated for children 16-30 months old.
Diagnostic Test: The Autism Spectrum Quotient Questionnaire -Children's Version — The Autism Spectrum Quotient-Children's Version (AQ-Child; Auyeung, Baron-Cohen, Wheelwright & Allison, 2008) is a parent report questionnaire that aims to quantify autistic traits in children 4 - 11 years old. It contains 50 likert-type items with responses ranging from "definitely agree" to "definitely disagree".
Diagnostic Test: The Autism-Spectrum Quotient (AQ)-Adolescent Version — The Autism Spectrum Quotient-Children's Version (AQ-Child; Auyeung, Baron-Cohen, Wheelwright & Allison, 2008) is a parent report questionnaire that aims to quantify autistic traits in children 12 - 15 years old. It contains 50 likert-type items with responses ranging from "definitely agree" to "definitely disagree".
Diagnostic Test: Continuous Movement Monitoring (Actimyo/Syde) — Continuous movement data will be collected using the ActiMyo/Syde® device (Servais et al., 2022), which is attached to the ankles and uses magneto-inertial sensors to quantify movement. At the first study visit, 20 ambulant patients older than 2 years old will be fitted with a Syde device to each ankle and their carers will be provided with training on use and care of the device. It will be worn for 30 days and then repeated in one year.
Diagnostic Test: Sleep Disturbance Scale for Children — The Sleep Disturbance Scale for Children (SDSC; Bruni et al., 1996) is a parent report questionnaire used to identify sleep disorders in children. It contains 26 likert-type items with responses ranging from "never" to "always (daily)". The items are divided in six categories - disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal/nightmares, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis (nighttime sweating).
Diagnostic Test: Seizure Diary — A 28-day seizure diary is a self-reported tool used to record seizure activity to obtain insight into the patient's seizure triggers and severity, monitor medication side effects, and promote medication adherence. Patients are asked to record their seizure occurrence, duration, and type of seizures.
Diagnostic Test: 30min EEG Recording — Recording will take place in the hospital's EEG department in a quiet room with low-light levels. If children will be unable to lay still, melatonin or dexmedetomidine may be used, as per standard department protocol. An EEG cap with international system 10-20 electrodes, ECG and respiratory electrodes will be placed on the head and chest respectively. Data will be recorded for at least 30 minutes, and an attempt will be made to capture both wakefulness and sleep. Intermittent photic stimulation will be performed as per standard protocol.
Diagnostic Test: PedsQL Family Impact Module — The PedsQL Family Impact Module is a parent report standardized questionnaire designed to measure the impact of paediatric chronic health conditions on the health-related quality of life (HRQOL) of parents and the functioning of the family as a whole. It consists of 36 likert-like items over 8 domains (Physical Functioning, Emotional Functioning, Social Functioning, Cognitive Functioning, Communication, Worry, Daily Activities, Family Relationships). The items are scored with responses ranging from "never a problem" to "always a problem".
Diagnostic Test: PedsQL Core Module — The PedsQL™ (Pediatric Quality of Life Inventory) Core Module is a health-related quality of life (HRQOL) questionnaire designed for children and adolescents. It assesses physical, emotional, social, and school functioning by using 23 likert-like items across 4 subscales (Physical Functioning, Emotional Functioning, Social Functioning, School Functioning). The items are scored with responses ranging from "never a problem" to "always a problem". Items differ across age groups - toddlers (2-4 years), young children (5-7 years), children (8-12 years), teens (13-18 years), and young adults (18-25 years). In toddlers, the parents serve as proxy, and in young children, a three-point scale with faces is used instead of likert-type responses.
Diagnostic Test: Blood Sample Collection — Venepuncture will be performed by a qualified member of the research team on all participants at each visit and 2x 5ml of blood will be collected (< 0.8 ml/kg) for analysis of DNA methylation and RNA expression, and analysis of serum for neurofilaments, b-catenin, and zinc. All blood samples will be labelled with the study ID and visit number and processed at the laboratory of the UMCL following the protocol "CTNNB1".
Diagnostic Test: Optical Coherence Tomography — To test for FEVR, the participants will be asked to perform Optical Coherence Tomography in their home countries at baseline and before or after every subsequent visit. OCT will only be performed in patients who will be able to cooperate - focus gaze for about 5 seconds.
Diagnostic Test: Brain MRI — If a participant has had a brain MRI performed prior to enrolling in our study, pictorial data will be analysed. If the participant will plan to have an MRI performed as a standard procedure in their native country, they will be asked to follow the CTNNB1 MRI protocol: T1 MPRAGE sequence, 3D FLAIR sequence, T2 axial planeartane, SWI, DWI, and DTI with at least 64, but preferably 90 diffusion directions. MRI will not be performed on site.

SUMMARY:
The aim of the Dragonfly study is to characterise and monitor the neurodevelopment of children and adults diagnosed with CTNNB1 syndrome through an international collaborative effort. Gaining comprehensive understanding of the mental, physical and social development of people with CTNNB1 neurodevelopmental syndrome and how their symptoms and abilities change over time will help improve and standardize care for these patients, as well as facilitate future research and clinical trials design.

DETAILED DESCRIPTION:
CTNNB1 syndrome is a rare debilitating neurodevelopmental disorder caused by mutations in the CTNNB1 gene, which is characterised by developmental delay and intellectual disability. Due to its relatively recent discovery, very little is known about the natural history of the condition. The aim of the Dragonfly study is to characterise and monitor the neurodevelopment of children and adults diagnosed with CTNNB1 syndrome through an international collaborative effort. This study is being conducted across several countries, including Slovenia, Spain, Brazil, the USA, and Australia.

In this natural history study, tinvestigators aim to recruit 150 children or adults of any age and phenotype with a confirmed genetic diagnosis of CTNNB1 syndrome, and their primary carers. Investigators will invite the participant and their carers to attend an annual study visit over a period of 5 years, during which investigators will collect retrospective and prospective clinical data. This will include a clinical neurological examination and assessments of motor and cognitive function, communication, behaviour, vision, sleep, assessment of gait using actimetry, and recordings of brain activity using electroencephalography (EEG). Investigators will also assess results of retinal assessment using Optical Coherence Tomography, and structural brain assessments using magnetic resonance imaging (MRI) - these diagnostic procedures will be performed in the participant's home county and not on site. Blood tests will be performed to reconfirm the underlying mutations in the CTNNB1 gene and investigate biomarkers of the condition. Carers will also be invited to complete questionnaires exploring their child's/dependent's abilities and the impact of the condition on their family's quality of life.

There is currently no curative treatment available for CTNNB1 syndrome. However, pre-clinical studies have been successfully completed with promising results and genetic therapies are currently in development. A comprehensive understanding of the natural progression of the condition is essential prior to commencing clinical trials of potential treatments. By improving our understanding of CTNNB1 syndrome, this study aims to lay the foundation for future clinical trials and the development of targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and genetically confirmed diagnosis of CTNNB1 syndrome.
* Age 0-99 years.
* Written informed consent/online consent to participate in study from a primary carer (parent or legal guardian).

Exclusion Criteria:

* Child/adult with CTNNB1 syndrome participating in a clinical trial of a potential treatment for the syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll individuals with a genetically confirmed pathogenic variant in the CTNNB1 gene consistent with a diagnosis of CTNNB1 neurodevelopmental syndrome. Each participant must have at least one parent or legal guardian available to support participation in the study. Families with more than one affected individual are eligible, and multiple participants from the same family may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Collection of relevant retrospective and prospective clinical data in patients with CTNNB1 syndrome via physical assessments, scales, and questionnaires. | 5 years
  The aim of the Dragonfly study is to characterise and monitor the neurodevelopment of children and adults diagnosed with CTNNB1 syndrome through an international collaborative effort. Gaining comprehensive understanding of the mental, physical and social development of people with CTNNB1 neurodevelopmental syndrome and how their symptoms and abilities change over time will help improve and standardize care for these patients, as well as facilitate future research and clinical trials design.

CONTACTS AND LOCATIONS:
Locations (2):
- Sydney Children's Hospital, Sydney, Australia
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakelj N, Gosar D, Mirosevic S, Sanders SJ, Ljungdahl A, Kohani S, Huang S, Leong LI, An Y, Teo MJ, Moultrie F, Jerala R, Lainscek D, Forstneric V, Susjan P, Lisowski L, Perez-Iturralde A, Mrak JO, Chan HYE, Osredkar D. Genotypic, functional, and phenotypic characterization in CTNNB1 neurodevelopmental syndrome. HGG Adv. 2025 Oct 9;6(4):100483. doi: 10.1016/j.xhgg.2025.100483. Epub 2025 Jul 18. PMID 40684264
- [Background] Mirosevic S, Khandelwal S, Susjan P, Zakelj N, Gosar D, Forstneric V, Lainscek D, Jerala R, Osredkar D. Correlation between Phenotype and Genotype in CTNNB1 Syndrome: A Systematic Review of the Literature. Int J Mol Sci. 2022 Oct 19;23(20):12564. doi: 10.3390/ijms232012564. PMID 36293418